CLINICAL TRIAL: NCT07392047
Title: Comparison Of The Efficacy Of 2% Metronidazole Gel Versus 1% Clindamycin Gel In The Treatment Of Moderate Acne Vulgaris
Brief Title: Metronidazole 2% Gel Versus Clindamycin 1% Gel for Moderate Acne Vulgaris
Acronym: METROCLIN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Rubab Murtaza, FCPS Resident, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JPMC-ACNE-RCT-01
Record Dates: First submitted 2026-01-27; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Acne Vulgaris
Keywords: Moderate acne; Metronidazole gel; Clindamycin gel; Topical antibiotic; Modified Global Acne Grading System
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Parallel-group, two-arm randomized controlled trial. Eligible participants with moderate acne vulgaris will be randomized in a 1:1 ratio using blocked randomization to receive either 2% metronidazole gel or 1% clindamycin gel, applied twice daily for 12 weeks, with follow-up assessments at weeks 4, 8, and 12.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronidazole 2% Gel (Experimental): Participants will apply 2% metronidazole gel as a thin layer twice daily (morning and night) for 12 weeks after gentle cleansing and drying.
  Interventions: Drug: Metronidazole Topical Gel 2%
- Clindamycin 1% Gel (Active Comparator): Participants will apply 1% clindamycin gel as a thin layer twice daily (morning and night) for 12 weeks after gentle cleansing and drying.
  Interventions: Drug: Clindamycin Topical Gel 1%

INTERVENTIONS:
Drug: Metronidazole Topical Gel 2% — Topical metronidazole gel 2% applied as a thin layer to affected areas twice daily (morning and night) for 12 weeks after gentle cleansing and drying.
  Arms: Metronidazole 2% Gel
Drug: Clindamycin Topical Gel 1% — Topical clindamycin gel 1% applied as a thin layer to affected areas twice daily (morning and night) for 12 weeks after gentle cleansing and drying.
  Arms: Clindamycin 1% Gel

SUMMARY:
Acne vulgaris is a common inflammatory skin disorder. This randomized controlled trial (RCT) will compare the efficacy and safety of 2% metronidazole gel versus 1% clindamycin gel in adults with moderate acne vulgaris at Jinnah Postgraduate Medical Centre (JPMC), Karachi. Sixty eligible participants (18-35 years) will be enrolled using consecutive sampling and randomized in a 1:1 ratio using blocked randomization. Participants will apply the assigned gel as a thin layer twice daily for 12 weeks. Acne severity will be assessed using the Modified Global Acne Grading System (mGAGS) at baseline and at weeks 4, 8, and 12. The primary outcome is the proportion of participants achieving at least a 50% reduction from baseline in total mGAGS score at week 12. Local adverse effects (e.g., erythema, itching, irritation) will be recorded at each follow-up visit.

DETAILED DESCRIPTION:
This is an investigator-initiated, parallel-group randomized controlled trial (RCT) conducted in the Department of Dermatology, Jinnah Postgraduate Medical Centre (JPMC), Karachi. After approval from the Institutional Review Board (IRB) and the College of Physicians and Surgeons Pakistan (CPSP), adults aged 18-35 years with moderate acne vulgaris, defined by a Modified Global Acne Grading System (mGAGS) score of 45-80, and not using other anti-acne therapies will be enrolled using non-probability consecutive sampling. Participants who are pregnant or lactating, have severe acne (mGAGS >80), have a known allergy to metronidazole or clindamycin, or have other dermatologic conditions affecting the face will be excluded.

Participants will be randomized in a 1:1 allocation using blocked randomization to receive either metronidazole 2% gel or clindamycin 1% gel. The assigned treatment will be applied as a thin layer twice daily (morning and night) for 12 weeks after gentle cleansing and drying of the face. Concomitant anti-acne products will be discouraged during the intervention period. Follow-up assessments will occur at weeks 4, 8, and 12. At each visit, acne severity will be assessed using mGAGS, and tolerability will be evaluated by recording local adverse effects, including erythema, itching, dryness, burning, or irritation.

The primary endpoint is treatment response at week 12, defined as a ≥50% reduction in total mGAGS score from baseline. Participants will be classified as responders (≥50% reduction) or non-responders (<50% reduction). Data will be analyzed using Statistical Package for the Social Sciences (SPSS) version 26. Categorical outcomes will be compared using the chi-square test or Fisher's exact test, and continuous variables will be compared using the independent-samples t test or Mann-Whitney U test according to data distribution. Stratified analyses will explore effect modification by age and sex. A two-sided p value ≤0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria

Adults aged 18-35 years of either sex.

Clinical diagnosis of moderate acne vulgaris, defined as a Modified Global Acne Grading System (mGAGS) score of 45-80.

Not currently using any other anti-acne treatment (topical or systemic).

Exclusion Criteria

Pregnant or lactating women.

Severe acne vulgaris, defined as an mGAGS score >80.

Known hypersensitivity/allergy to metronidazole or clindamycin (or any component of the study gels).

Any other dermatologic condition affecting the face that may interfere with assessment of acne severity or treatment response.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Treatment response by mGAGS at Week 12 | 12 weeks
  Proportion of participants achieving ≥50% reduction in total Modified Global Acne Grading System (mGAGS) score from baseline (Responder = Yes; Non-responder = No).

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the study team. Data will be stored securely at the study site and used only for the purposes described in the protocol. Aggregate, de-identified results will be reported in publications

REFERENCES:
- [Result] 20. Verma R, Yadav P, Chudhari M, Patel J, Umrigar D. Comparison of efficacy of two topical drug therapy of acne vulgaris-1% clindamycin versus 5% dapsone: a split-face comparative study. Natl J Physiol Pharm Pharmacol. 2022;12(6):817-822.
- [Result] 19. Irshad M, Syed AW, Shah MW, Naeem U, Mirza M, Naeem S. Comparative effects of azithromycin and probiotics for treatment of acne vulgaris. J Coll Physicians Surg Pak. 2023;33(5):516-520.
- [Result] 18. Naveed S, Masood S, Rahman A, Awan S, Tabassum S. Impact of acne on quality of life in young Pakistani adults and its relationship with severity: a multicenter study. Pak J Med Sci. 2021;37(3):727-732. doi:10.12669/pjms.37.3.2819
- [Result] 17. Dessinioti C, Katsambas A. Antibiotics and antimicrobial resistance in acne: epidemiological trends and clinical practice considerations. Yale J Biol Med. 2022;95(1):53-63.
- [Result] 16. Dréno B, Corvec S, et al. Acne microbiome: From phyla to phylotypes. J Eur Acad Dermatol Venereol. 2024;38(4):657-664. doi:10.1111/jdv.19540
- [Result] 15. Chen X, et al. Metronidazole: the clinical efficacy and pharmacological effects. Biomedicines. 2023;11(8):2153. doi:10.3390/biomedicines11082153
- [Result] 14. Khodaeiani E, Fouladi RF, Yousefi N, Amirnia M, Babaeinejad S, Shokri J. Efficacy of 2% metronidazole gel in moderate acne vulgaris. Indian J Dermatol. 2012;57(4):279-281. doi:10.4103/0019-5154.97666
- [Result] 13. Nakase K, Aoki S, Sei S, Fukumoto S, Horiuchi Y, Yasuda T, et al. Characterization of acne patients carrying clindamycin-resistant Cutibacterium acnes: a Japanese multicenter study. J Dermatol. 2020;47(8):863-869. doi:10.1111/1346-8138.15397
- [Result] 12. Aoki S, Nakase K, Nakaminami H, Wajima T, Hayashi N, Noguchi N. Transferable multidrug-resistance plasmid carrying a novel macrolide-clindamycin resistance gene, erm(50), in Cutibacterium acnes. Antimicrob Agents Chemother. 2020;64(3):e01810-19. doi:10.1128/AAC.01810-19
- [Result] 11. Koyanagi S, Koizumi J, Nakase K, Hayashi N, Horiuchi Y, Watanabe K, et al. Increased frequency of clindamycin-resistant Cutibacterium acnes strains isolated from Japanese patients with acne vulgaris caused by the prevalence of exogenous resistance genes. J Dermatol. 2023;50(6):793-799. doi:10.1111/1346-8138.16757
- [Result] 10. Beig M, et al. Prevalence of antibiotic-resistant Cutibacterium acnes isolated from acne patients: a systematic review and meta-analysis. Lancet Reg Health Southeast Asia. 2024. doi:10.1016/j.lansea.2024.100137
- [Result] 9. American Academy of Dermatology. Guidelines of care for the management of acne vulgaris. J Am Acad Dermatol. 2024. doi:10.1016/j.jaad.2023.12.017
- [Result] 8. Khodaeiani E, Fouladi RF, Yousefi N, Amirnia M, Babaeinejad S, Shokri J. Efficacy of 2% metronidazole gel in moderate acne vulgaris. Indian J Dermatol. 2012;57(4):279-81.
- [Result] 7. Verma R, Yadav P, Chudhari M, Patel J, Umrigar D. Comparison of efficacy of two topical drug therapy of acne vulgaris - 1% clindamycin versus 5% dapsone: A split face comparative study. Natl J Physiol Pharm Pharmacol. 2022;12(6):817-22
- [Result] 6. Rahim S, Kumar A. The impact of acne vulgaris on quality of life and psychic health in young adolescents of Rehman Medical College, Peshawar, Pakistan: a cross-sectional study. J Rehman Med Inst. 2024;8(1):1-5.
- [Result] 5. Babar O, Mobeen A. Prevalence and psychological impact of acne vulgaris in female undergraduate medical students of Rawalpindi and Islamabad, Pakistan. Cureus. 2019;11(10)
- [Result] 4. Irshad M, Syed AW, Shah MW, Naeem U, Mirza M, Naeem S. Comparative effects of azithromycin and probiotics for treatment of acne vulgaris. J Coll Physicians Surg Pak. 2023;33(5):516-20.
- [Result] 3. Rahim S, Kumar A. The impact of acne vulgaris on quality of life and psychic health in young adolescents of Rehman Medical College, Peshawar, Pakistan: a cross-sectional study. J Rehman Med Inst. 2024;8(1):1-5
- [Result] 2. Babar O, Mobeen A. Prevalence and psychological impact of acne vulgaris in female undergraduate medical students of Rawalpindi and Islamabad, Pakistan. Cureus. 2019;11(10)
- [Result] 1. Irshad M, Syed AW, Shah MW, Naeem U, Mirza M, Naeem S. Comparative effects of azithromycin and probiotics for treatment of acne vulgaris. J Coll Physicians Surg Pak. 2023;33(5):516-20.